CLINICAL TRIAL: NCT00414154
Title: The Effect of a Group Based Multidisciplinary Patient Education Programme for Patients With Osteoporosis - a Controlled Randomised Trial
Brief Title: The Importance of Patient Education - A Randomised Controlled Trial
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 026
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2007-03

CONDITIONS: Osteoporosis; Quality of Life; Level of Adherence; Behavior
Keywords: Group based patient education,; multidisciplinary,; physical activity,; adherence to treatment,; quality of life
MeSH Terms: conditions — Osteoporosis; Behavior; Motor Activity; Treatment Adherence and Compliance

INTERVENTIONS:
Behavioral: Group based multidisciplinary patient education programme

SUMMARY:
Modification of individual life style factors and fall prevention programmes may have significant positive effects on fracture incidence. Also, a large number of studies have demonstrated that pharmacological therapy of osteoporosis is effective; however non-adherence to such therapy is a well recognized problem. Few studies, however, have examined the effect of particular patient education programmes on knowledge and adherence to therapy.

We hypothesised that a group-based, multi-disciplinary, education programme increases the total quality of treatment for patients with osteoporosis, Patients' knowledge on osteoporosis and adherence with pharmacological therapy ect.

A total of 300 patients, recently diagnosed with osteoporosis and started on specific treatment, were randomised to either the "school" or "control" group. In the school-group, patients attended four classes with 8-12 participants during four weeks (a total of 12 hours). Teaching was performed by nurses, physiotherapists, dieticians, and doctors and was based on dialogs and situated learning. The classes covered "facts on osteoporosis", "fractures and pain", "diet", "preventive measures", "balance and exercise", and "medical treatment". Teaching was designed to increase empowerment. The control group were offered the department's standard treatment including follow-up visits.

All 300 patients received questionnaires regarding "Knowledge about Osteoporosis", "Level of Adherence", "Quality of life", "Dietary calcium intake", "Level of physical activity", "Falls events" registered every month by postcard, at inclusion and after 3, 12, and 24 month. BMD was examined by DXA-scan at inclusion and after 12 and 24 month. The last patient will answer the questionnaires first of May 2007.

ELIGIBILITY:
Inclusion Criteria:

* Men and female age 45-80,
* Diagnosed with osteoporosis and started medical treatment

Exclusion Criteria:

* Severe illness,
* Cognitive dysfunction,
* Not able to speak or read Danish

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-05; Study Completion 2007-05

PRIMARY OUTCOMES:
Level of compliance to pharmacological treatment

SECONDARY OUTCOMES:
Quality of life,
Level of physical activity,
Daily dietary calcium intake,
registration of fall in and outdoor,
Knowledge on Osteoporosis, BMD

CONTACTS AND LOCATIONS:
Overall Officials: Kim Brixen, MD, Ph.D, Principal Investigator — Institute of Clinical Research, University of Southern Denmark
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Odense, Denmark